CLINICAL TRIAL: NCT01241669
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of Multiple Doses of E5555 on the Pharmacokinetics of Metformin (a Substrate for OCT2 Transporter) and on Renal Function in Healthy Subjects
Brief Title: Randomized, Placebo-controlled Study to Evaluate Effects of E5555 on Renal Function Parameters and OCT2 Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E5555-A001-023
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — E 5555

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: E5555
- Arm 2 (Experimental)
  Interventions: Drug: E5555

INTERVENTIONS:
Drug: E5555 — Drug: Oral E5555 400 mg/matching placebo, oral metformin 500 mg, iohexal 20 mL intravenous (IV), and para-aminohippuric acid (PAH) 7 mg/kg IV.
  Arms: Arm 1
Drug: E5555 — Drug: Oral E5555 100 mg/matching placebo, oral metformin 500 mg, iohexal 20 mL intravenous (IV), and para-aminohippuric acid (PAH) 7 mg/kg IV bolus.
  Arms: Arm 2

SUMMARY:
This is a drug-drug interaction study to evaluate the effects of steady-state exposure of E5555 and its main metabolites on the pharmacokinetics (PK) of metformin, an organic cation transporter-2 (OCT2) substrate. In addition, the study will also investigate the effects of E5555 on several renal function parameters.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male or female subjects aged greater than or equal to 18 years to 55 years

Exclusion Criteria:

* History of any medical condition which will result in an increased risk of bleeding including but not limited to active or recurrent gastric ulcers, recent head trauma or surgery, severe hypertension, bacterial endocarditis, etc.
* Creatinine clearance < 90 mL/min as estimated using Cockcroft-Gault formula at screening or baseline
* History of any renal disorders, proteinuria, hepato-biliary disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of multiple doses of E5555 on single dose pharmacokinetics of metformin. | 15 days

SECONDARY OUTCOMES:
To assess the effects of multiple doses of E5555 on the glomerular filtration rate estimated using iohexol. | Days 7 and 14
To assess the effects of multiple doses of E5555 on the effective renal plasma flow estimated using para-aminohippuric acid (PAH). | Days 7 and 14
To assess the multiple dose pharmacokinetics of E5555 and its main 6 metabolites. | Days 12-18
To assess the safety and tolerability of multiple doses of E5555 and a single dose of metformin either given alone or concomitantly | Day 1 - Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Bhaskar Rege, Study Director — Eisai Inc.
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States